CLINICAL TRIAL: NCT00024661
Title: Study to Determine the Maximum Tolerated Dose of Liposome-Encapsulated C-RAF Antisense Oligodeoxynucleotide (LErafAON) in Patients With Advanced Solid Tumors
Brief Title: Study to Determine the Maximum Tolerated Dose of LErafAON in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Collaborators: Georgetown University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LErafAON-002
Record Dates: First submitted 2001-09-24; First posted 2001-09-25 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Neoplasms
Keywords: recurrent solid tumors; liposomes containing AON to c-raf protein (LErafAON)
MeSH Terms: conditions — Neoplasms | interventions — LErafAON

INTERVENTIONS:
Drug: LErafAON

SUMMARY:
LErafAON is a liposome encapsulated c-raf antisense oligonucleotide. Raf-1 is a protein produced by human cells, both normal and cancerous, which may help protect tumor cells from radiation. Antisense oligonucleotides are very specific drugs, which can decrease the amount of a certain target protein by blocking the gene that makes it. Antisense oligonucleotide to raf gene can reduce the amount of Raf-1 protein in tumor cells. Liposomes are tiny globules of fat, which can carry drugs in the body. The experimental agent LErafAON is composed of liposomes carrying antisense oligonucleotide against the Raf-1 protein. It is hoped that decreased Raf-1 in the cancer cells will make them more sensitive to the radiation therapy.

Patients with advanced solid tumors will receive IV infusions of LErafAON over at least 60 minutes, once per week, for 8 weeks. In the absence of progression, patients may continue on weekly treatment. Pre-medications will be administered prior to each dose of study medication.

Cohorts of at least three patients will be entered at escalating dose-levels. Each cohort will be observed for at least ten days after receiving the first dose of treatment before additional patients are treated at a higher dose level. Patients will be followed for one month after receiving the last dose of study medication. The study will stop when a maximum tolerated dose (MTD) is identified. Dose escalation within a patient will not be allowed.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and MTD of LErafAON when given by weekly IV infusion for 8 weeks in patients with advanced malignancies.

II. Characterize the plasma pharmacokinetics of LErafAON after IV infusion.

III. Document in vivo inhibition of Raf-1 protein by LErafAON.

IV. Detect anti-tumor effects of intravenous LErafAON.

PROTOCOL OUTLINE: This is a Phase I Maximum Tolerated Dose (MTD) study for patients with recurrent solid tumor malignancies. Study medication will be administered by intravenous infusion over at least 60 minutes, once per week, for 8 weeks. In the absence of progression, patients may continue on weekly treatment. Pre-medications will be administered prior to each dose of study medication. Patients will be followed for one month after receiving the last dose of study medication. Patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) at the Week 8 disease assessment may continue to receive study medication until disease progression (PD).

Cohorts of at least three patients will be entered at escalating dose-levels. Each cohort will be observed for at least ten days after receiving the first dose of treatment before additional patients are treated at a higher dose level. Patients will be followed for one month after receiving the last dose of study medication. The study will stop when a maximum tolerated dose (MTD) is identified. Dose escalation within a patient will not be allowed.

PROJECTED ACCRUAL: Estimated enrollment is 15-35 patients; 3 per dose level, expanded to 6 if DLT occurs.

ELIGIBILITY:
-Disease Characteristics-

Histologically-confirmed malignancy which has recurred or progressed after initial definitive treatment and/or for which no curative therapy is available.

At least 30 days must have elapsed since receiving an investigational agent, at least 21 days since receiving any prior chemotherapy, and at least six weeks since receiving nitrosourea-containing therapy; patient must have recovered from any related side effects.

Must have a measurable or evaluable tumor documented within 4 weeks prior to having study-related procedures.

-Patient Characteristics-

Performance Status (ECOG) of 0 - 2.

Must be at least 18 years of age.

Must have adequate organ function: Absolute neutrophil count at least 1,500/mm3; Platelets at least 100,000/mm3; Creatinine, Calcium, and total Bilirubin not higher than the upper limit of normal; Liver enzymes AST and ALT not more than 2.5 x the upper limit of normal; PT and aPTT not more than the upper limit of normal.

Life expectancy more than 12 weeks.

Must sign Informed Consent.

No concurrent antitumor therapy.

No infection requiring parenteral antibiotics; no HIV infection; no chronic hepatic disease; and no seropositivity for Hepatitis B and Hepatitis C. (Use of prophylactic antibiotics is permitted.)

No pregnant or lactating females. All females of child-bearing potential must use an effective method of contraception.

No active Central Nervous System (CNS) metastasis. Neuroimaging is required only if metastasis is suggested by history or physical examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2001-03; Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Charles Rudin, M.D., Principal Investigator
Locations (3):
- United States (3):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Temple University Cancer Center, Philadelphia, Pennsylvania